CLINICAL TRIAL: NCT02108288
Title: Pharmacokinetic Study of OPC-1085EL Ophthalmic Solution in Healthy Male Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1085EL-13-004
Record Dates: First submitted 2014-03-27; First posted 2014-04-09 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OPC-1085EL ophthalmic solution (Experimental): Once daily
  Interventions: Drug: OPC-1085EL ophthalmic solution
- Carteolol long-acting ophthalmic solution (Active Comparator): Once daily
  Interventions: Drug: Carteolol long-acting ophthalmic solution
- Latanoprost ophthalmic solution (Active Comparator): Once daily
  Interventions: Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: OPC-1085EL ophthalmic solution
  Arms: OPC-1085EL ophthalmic solution
Drug: Carteolol long-acting ophthalmic solution
  Arms: Carteolol long-acting ophthalmic solution
Drug: Latanoprost ophthalmic solution
  Arms: Latanoprost ophthalmic solution

SUMMARY:
OPC-1085EL ophthalmic solution, carteolol long-acting ophthalmic solution or latanoprost ophthalmic solution are administered once daily for 7 days and the effect on the blood concentration of carteolol and latanoprost in OPC-1085EL ophthalmic solution by formulating the combination drug will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are considered medically healthy per investigator's judgment

Exclusion Criteria:

* Subjects with ocular conditions as defined by the protocol
* Subjects with intraocular pressure: <10 or ≥22 mmHg

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kansai Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-1085EL Ophthalmic Solution: Once daily
  OPC-1085EL ophthalmic solution
- Carteolol Long-acting Ophthalmic Solution: Once daily
  Carteolol long-acting ophthalmic solution
- Latanoprost Ophthalmic Solution: Once daily
  Latanoprost ophthalmic solution
Period: Overall Study
Arm/Group | OPC-1085EL Ophthalmic Solution | Carteolol Long-acting Ophthalmic Solution | Latanoprost Ophthalmic Solution
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-1085EL Ophthalmic Solution | Carteolol Long-acting Ophthalmic Solution | Latanoprost Ophthalmic Solution | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (5.7) | 25.5 (3.0) | 24.0 (2.8) | 25.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  Japan | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Carteolol
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OPC-1085EL Ophthalmic Solution | Carteolol Long-acting Ophthalmic Solution
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 1 | 0.8558 (0.2658) | 0.9984 (0.4832)
  Day 7 | 1.174 (0.3085) | 1.627 (0.5001)

2. Primary Outcome: Cmax of Latanoprost Acid
Time Frame: Day 1 and Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 10 | 10
pg/mL
  Day 1 | 19.77 (10.13) | 21.22 (10.16)
  Day 7 | 18.47 (8.913) | 17.48 (8.892)

3. Secondary Outcome: Tmax of Carteolol
Time Frame: Day 1 and Day 7
Measure: Median (Full Range); unit: h
Arm/Group | OPC-1085EL Ophthalmic Solution | Carteolol Long-acting Ophthalmic Solution
Number analyzed (Participants) | 10 | 10
h
  Day 1 | 0.25 [0.25 to 4.00] | 0.25 [0.25 to 23.92]
  Day 7 | 0.25 [0.25 to 4.00] | 0.38 [0.25 to 24.00]

4. Secondary Outcome: Tmax of Latanoprost Acid
Time Frame: Day 1 and Day 7
Measure: Median (Full Range); unit: min
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 10 | 10
min
  Day 1 | 10 [5 to 10] | 10 [5 to 10]
  Day 7 | 5 [5 to 10] | 10 [5 to 10]

ADVERSE EVENTS:
Time Frame: Up to 24 days from date of informed consent
Arm/Group | OPC-1085EL Ophthalmic Solution | Carteolol Long-acting Ophthalmic Solution | Latanoprost Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 4/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-1085EL Ophthalmic Solution (N=10) | Carteolol Long-acting Ophthalmic Solution (N=10) | Latanoprost Ophthalmic Solution (N=10)
Accommodation disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 6 (10) | 3 (3) | 8 (11)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No